CLINICAL TRIAL: NCT05224661
Title: Molecular Evaluation of AML Patients After Stem Cell Transplant to Understand Relapse Events
Acronym: MEASURE
Status: Active, not recruiting | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other)
Responsible Party: Sponsor
Other Study IDs: MEASURE
Record Dates: First submitted 2021-11-22; First posted 2022-02-04 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia in Remission

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Bone Marrow (if collected for clinical purposes only), archived specimens from time of AML diagnosis (diagnosis specimens include: bone marrow aspirate cells, extracted DNA, marrow aspirate pellet, marrow aspirate slides, blood)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with AML in complete remission undergoing alloHCT: Adult patients with AML in complete remission undergoing alloHCT
  Interventions: Other: Prospective determination of the clinical utility of measurable residual disease (MRD) testing

INTERVENTIONS:
Other: Prospective determination of the clinical utility of measurable residual disease (MRD) testing — Prospective determination of the clinical utility of measurable residual disease (MRD) testing for relapse and survival of patients with acute myeloid leukemia (AML) undergoing allogeneic hematopoietic cell transplantation (alloHCT).

SUMMARY:
Prospective determination of the clinical utility of measurable residual disease (MRD) testing for relapse and survival of patients with acute myeloid leukemia (AML) undergoing allogeneic hematopoietic cell transplantation (alloHCT).

DETAILED DESCRIPTION:
This is a multi-center non-randomized prospective study designed to establish a national framework for introducing measurable residual disease testing into the clinical care of AML patients undergoing allogeneic transplantation.

Enrollment is expected to occur over a 4-year period, with an additional 3 years of follow-up. Subject participation this study will be approximately 3 years. Up to 1,000 subjects will be enrolled.

Subjects will be asked to provide blood samples at months 1-6, 9, 12, 15, and 18 post-transplant, and archived specimens from time of AML diagnosis and any bone marrow samples collected for clinical purposes will be requested for research testing. Additional blood and marrow samples will be requested at relapse (if applicable).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Aged at least 18 years old at time of consent
4. Diagnosed with AML, in complete remission

   1. Complete remission (CR) definition per local institutional criteria
   2. CR with incomplete hematologic recovery (CRi) is not an exclusion criterion
   3. MRD positivity is not an exclusion criterion
5. Undergoing alloHCT
6. Has a diagnostic AML specimen available

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia
2. Prior alloHCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with AML in complete remission undergoing alloHCT
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Through up to 3 years post-alloHCT
  Overall survival post-alloHCT via comparison between those testing positive or negative using an optimized molecular monitoring approach.
Cumulative incidence of relapse | Through up to 3 years post-alloHCT
  Cumulative incidence of relapse post-alloHCT via comparison between those testing positive or negative using an optimized molecular monitoring approach.

SECONDARY OUTCOMES:
Relapse Prediction - Testing Approaches | Through up to 3 years post-alloHCT
  Proportion of post-alloHCT relapses identified by different MRD testing approaches with optimal test thresholds at peri-transplant timepoints.
Relapse Prediction - Pre-Transplant Testing | Through up to 3 years post-alloHCT
  Proportion of post-alloHCT relapses predicted by pre-transplant testing (comparing blood with marrow when available).
Relapse Prediction - Early Prediction | Through up to 3 years post-alloHCT
  Proportion of post-alloHCT relapses identified one month or more earlier than local testing by post-alloHCT optimized monitoring.
Relapse Prediction - Time to Relapse | Through up to 3 years post-alloHCT
  Time from testing positive by optimized monitoring to relapse.
Biology of Relapse - Change in Genetic Profile | Through up to 3 years post-alloHCT
  for subjects with relapse sample available) - Proportion of relapses with change in genetic profile to diagnosis.
Biology of Relapse - Change in Immunophenotype | Through up to 3 years post-alloHCT
  (for subjects with relapse sample available) - Proportion of relapses with change in immunophenotype to diagnosis.
Biology of Relapse - HLA Loss | Through up to 3 years post-alloHCT
  (for subjects with relapse sample available) - Proportion of relapses with evidence of human leukocyte antigen (HLA) loss.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hourigan, DM, D.Phil., Study Chair — Virginia Polytechnic Institute and State University; Jeffrey Auletta, MD, Study Chair — National Marrow Donor Program
Locations (18):
- United States (18):
  - City of Hope, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian / Weill Cornell Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Fred Hutchinson Cancer Center, Seattle, Washington

DOCUMENTS (1):
  • Informed Consent Form (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT05224661/ICF_000.pdf